CLINICAL TRIAL: NCT02984813
Title: Measurement of Oxidative Stress of Retinal Ganglion Cells With and Without Anti-oxidants and Anti-inflammatory Agents in Patients With Glaucoma and Diabetic Retinopathy as Determined by Mitochondrial Flavoprotein Fluorescence
Brief Title: Safety and Efficacy of Anti-Oxidants and Anti-inflammatory Agents in Glaucoma and Diabetic Retinopathy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator left the institution
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15.25
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Open-angle Glaucoma; Diabetic Retinopathy
MeSH Terms: conditions — Glaucoma, Open-Angle; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GlaucoHealth (Experimental): 2 pills once daily in the morning for 3 months
  Interventions: Drug: GlaucoHealth
- GlaucoSelect (Experimental): 2 pills once daily in the morning for 3 months
  Interventions: Drug: GlaucoSelect
- Placebo (Placebo Comparator): 2 pills once daily in the morning for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GlaucoHealth — Containing alpha lipoic acid, citicoline, Co-enzyme Q10, Ginkgo biloba extract, grape seed extract, N-acetyl-cysteine, curcumin, and green tea extract
  Arms: GlaucoHealth
Drug: GlaucoSelect — Containing curcumin, bilberry extract, and grape seed extract
  Arms: GlaucoSelect
Drug: Placebo — No active ingredients
  Arms: Placebo

SUMMARY:
This study is a multi-armed protocol designed to evaluate the safety and efficacy of two different combinations of nutritional supplements (study drug) (Glauco-Health and Glauco-Select) chosen for their potential to protect retinal ganglion cells against oxidative stress, low-grade inflammation, and mitochondrial dysfunction in patients with open-angle glaucoma and diabetic retinopathy. Oxidative stress and retinal cellular dysfunction will be measured using a Retinal Metabolic Analyzer (RMA) in this randomized, single center, double masked study. Patients with glaucoma will be divided into three treatment arms randomized to receive either Glauco-Health, Glauco-Select, or placebo.

DETAILED DESCRIPTION:
This investigation is using over the counter supplements. The investigation is intended only to evaluate their effect on the structure or function of mitochondria as it relates to the autofluorescence imaging being conducted in the study. They are not being studied to evaluate their ability to diagnose, cure, mitigate, or treat disease.

These ingredients in these combinations of nutritional supplements have also been reported beneficial in diabetic retinopathy. Patients with diabetic retinopathy will be added later as an additional arm and an amendment to this effect will be submitted when that portion of the study is ready to be initiated. That amendment will include background material, appropriate inclusion and exclusion criteria, informed consent, and references. At the current time, only the glaucoma proposal and glaucoma patients will be enrolled according to this submitted protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race, at least 18 years of age.
2. Has provided verbal and written informed consent.
3. Able and willing to follow instructions, including participation in all study assessments and visits.
4. Eyes with moderate to severe primary open-angle glaucoma will be enrolled. Glaucoma severity will be graded using the WHO glaucoma staging system.

   1. OAG eyes are defined by clinical findings consistent with glaucomatous optic neuropathy (Ex: thinning, excavation, rim erosion or notching of the neuroretinal rim)
   2. Reproducible visual field defects on at least three examinations as measured by a glaucoma hemifield test (GHT) result outside normal limits and/or the presence of at least three consecutive test points on the pattern deviation plot with P<1% and at least one at P<0.05%, not including points on the edge of the field.
5. Both eyes will be enrolled.
6. Refractive error ≤5 diopters and astigmatism ≤3 diopters

Exclusion Criteria:

1. Comorbidity with other severe or chronic eye conditions that in the judgment of the investigator will interfere with study assignment, such as age-related macular degeneration, macular dystrophy, retinopathy from systemic diseases, marked ocular media opacities that obscure retinal imaging, etc.
2. BCVA <20/200
3. Concurrent conjunctivitis, keratitis or uveitis
4. History of penetrating ocular trauma.
5. Subject uncooperativeness that restricts adequate examination of IOP, ocular fundus or anterior chamber.
6. Has a condition or history that, in the opinion of the investigator, may interfere significantly with the subject's participation in the study.
7. A woman who is pregnant, nursing an infant, or planning a pregnancy
8. Has a known adverse reaction and/or sensitivity to the study drug or its compound.

   a. Including: alpha lipoic acid, citicoline, Co-enzyme Q-10, Ginkgo biloba extract, grape seed extract, N-acetyl-cysteine, curcumin, green tea extract, and bilberry extract.
9. Currently enrolled in an investigational drug study or has used an investigational drug within 30 days prior to Visit 1.
10. Is planning on having surgery at any time throughout the study duration (90 days from initiation)
11. Is currently receiving chemotherapy
12. Has a history of diabetes mellitus, seizure(s), bleeding disorder(s)
13. Has a history of uncontrolled hypertension (≥180 systolic or ≥110 diastolic on two successive measures)
14. Has a history of any radiation around the eyes
15. Currently using anticoagulant/antiplatelet drugs (patients on coumadin, clopidogral (Plavix), and plasugrel (Effient) will be excluded but that patients taking aspirin will be allowed)
16. Unwilling or unable to cease using other anti-oxidative agents or drugs.
17. Dilated pupil diameter less than 5 millimeters
18. Fluorescein drop administration within 8 hours before imaging
19. History of cataract surgery in the 3 months prior to imaging
20. History of any other intraocular surgery within 4 months prior to enrollment
21. Corticosteroid or immunosuppressive therapy within 6-months prior to imaging
22. Lens opacity ≥grade 3 on ARLNS on standard photographs (Appendix 6)
23. History of vitrectomy
24. Monocular patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Flavoprotein fluorescence index | 3 months
  Average Intensity and Average Curve Width

SECONDARY OUTCOMES:
Visual acuity | 3 months
Humphrey visual field testing (24-2) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ritch, MD, Principal Investigator — Shelley and Steven Einhorn Distinguished Chair Professor of Ophthalmology Surgeon Director Emeritus and Chief, Glaucoma Services The New York Eye and Ear Infirmary of Mount Sinai
Locations (1):
- New York Eye and Ear Infirmary of Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided